CLINICAL TRIAL: NCT02438436
Title: Influence of Simo Decoction Plus Acupuncture and Gum Chewing on Postoperative Bowel Activity After Resection for Patients With HCC
Brief Title: Simo Decoction and Gum Chewing for Bowel Activity
Acronym: SD/GC-HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Guangxi Medical University, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SD/GC-HCC
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- simo decoction (Experimental): Patients will receive simo decoction (10 mL/piece,three times per day) and bilateral tsusanli acupoint injections with vitamin B1 two times per day, starting in the first day after resection until flatus.
  Interventions: Dietary Supplement: simo decoction
- gum chewing (Active Comparator): Patients will receive gum chewing (three times per day) in the first day after resection until flatus.
  Interventions: Other: gum chewing
- empty control (No Intervention)

INTERVENTIONS:
Dietary Supplement: simo decoction
  Arms: simo decoction
Other: gum chewing
  Arms: gum chewing

SUMMARY:
Abdominal surgery, including hepatic resection for hepatocellular carcinoma (HCC), is inevitably followed by an episode of gastrointestinal hypomotility. A delayed return of gastrointestinal function, defined as postoperative ileus (POI), has a great impact on patient comfort, morbidity and recovery. POI often results in a prolonged hospital stay and contributes significantly to healthcare costs.

Some prospective studies have revealed that gum chewing can improve the return of gastrointestinal function after colorectum surgery, gynaecology and obstetrics, and urinary system surgery. Moreover, some retrospective studies also revealed that simo decoction may improve the return of gastrointestinal function after hepatic resection of HCC. Therefore, the present study compared the effect of gum chewing and simo decoction after hepatic resection of HCC on POI, surgical complications, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Underwent open hepatic resection
* Diagnosis of HCC was confirmed by histopathological examination of surgical samples in all patients

Exclusion Criteria:

* Previously underwent exploratory laparotomy
* Laparoscopic surgery
* Known Central Nervous System tumors including metastatic brain disease
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
First flatus time | one day
xerostomia | one day

CONTACTS AND LOCATIONS:
Overall Officials: Le-Qun Li, MD, Study Chair — Guangxi Medical University Cancer Hospital
Locations (1):
- Department of Hepatobilliary Surgery, Affiliated Tumor of Guangxi University, Nanning, Guangxi, China

REFERENCES:
- [Background] Jang SY, Ju EY, Kim DE, Kim JH, Kim YH, Son M, Jang M, Jeong JH, Kim KS. First flatus time and xerostomia associated with gum-chewing after liver resection. J Clin Nurs. 2012 Aug;21(15-16):2188-92. doi: 10.1111/j.1365-2702.2012.04132.x. Epub 2012 Jun 2. PMID 22672009
- [Background] van den Heijkant TC, Costes LM, van der Lee DG, Aerts B, Osinga-de Jong M, Rutten HR, Hulsewe KW, de Jonge WJ, Buurman WA, Luyer MD. Randomized clinical trial of the effect of gum chewing on postoperative ileus and inflammation in colorectal surgery. Br J Surg. 2015 Feb;102(3):202-11. doi: 10.1002/bjs.9691. Epub 2014 Dec 18. PMID 25524125
- [Result] You XM, Mo XS, Ma L, Zhong JH, Qin HG, Lu Z, Xiang BD, Wu FX, Zhao XH, Tang J, Pang YH, Chen J, Li LQ. Randomized Clinical Trial Comparing Efficacy of Simo Decoction and Acupuncture or Chewing Gum Alone on Postoperative Ileus in Patients With Hepatocellular Carcinoma After Hepatectomy. Medicine (Baltimore). 2015 Nov;94(45):e1968. doi: 10.1097/MD.0000000000001968. PMID 26559269
- See also: This study is completed. — https://journals.lww.com/md-journal/Fulltext/2015/11110/Randomized_Clinical_Trial_Comparing_Efficacy_of.24.aspx